CLINICAL TRIAL: NCT06524596
Title: Wuhan Children's Hospital
Brief Title: Study on Gynecological Laparoscopy Under Total Intravenous Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan Children's Hospital (Other)
Responsible Party: Principal Investigator, Xiang Wang, MM, Wuhan Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WHCH-008
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Butorphanol
Keywords: Analgesia; Remifentanil; Postoperative Pain
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Saline Solution; Propofol; Remifentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the butorphanol group (Experimental): 0.02 mg/kg of tartaric acid butorphanol intravenously 30 minutes prior to anaesthesia induction.
  Interventions: Drug: tartaric acid butorphanol; Drug: propofol and remifentanil
- the control group (Placebo Comparator): 0.02 mg/kg of normal saline intravenously 30 minutes prior to anaesthesia induction.
  Interventions: Drug: normal saline; Drug: propofol and remifentanil

INTERVENTIONS:
Drug: tartaric acid butorphanol — The group received 0.02 mg/kg tartaric acid butorphanol intravenously over 5 minutes, 30 minutes before anaesthesia induction
  Arms: the butorphanol group
Drug: normal saline — The group received 0.02 mg/kg normal saline intravenously over 5 minutes, 30 minutes before anaesthesia induction
  Arms: the control group
Drug: propofol and remifentanil — Anaesthesia was induced with 2 mg/kg propofol and 0.6 μg/kg remifentanil and maintained with a target-controlled infusion (TCI) of propofol and remifentanil, using the Marsh and Minto models, respectively.

SUMMARY:
To investigate the effect of preemptive analgesia with tartaric acid butorphanol on postoperative pain in gynecological laparoscopy under total intravenous anesthesia with remifentanil.This randomised, double-blind, placebo-controlled trial enrolled 60 patients undergoing elective gynaecological laparoscopy. The patients were divided into two groups: the butorphanol group (n = 30) and the control group (n = 29). Both groups received TIVA with propofol and remifentanil. Observing two groups of patients on the visual analog scale, the total consumption of rescue analogies, and the confidence of postoperative nausea and vomiting (PONV), and the patient satisfaction score.

DETAILED DESCRIPTION:
To investigate the effect of preemptive analgesia with tartaric acid butorphanol on postoperative pain in gynecological laparoscopy under total intravenous anesthesia with remifentanil.This randomised, double-blind, placebo-controlled trial enrolled 60 patients undergoing elective gynaecological laparoscopy. The patients were divided into two groups: the butorphanol group (n = 30), who received 0.02 mg/kg of tartaric acid butorphanol intravenously 30 minutes prior to anaesthesia induction, and the control group (n = 29), who received the same volume of normal saline. Both groups received TIVA with propofol and remifentanil. The primary outcome was the visual analogue scale (VAS) score for pain at rest and on movement at 1, 2, 4, 6, 12 and 24 hours after surgery. The secondary outcomes were the total consumption of rescue analgesics, the incidence and severity of postoperative nausea and vomiting (PONV), and the patient satisfaction score.

ELIGIBILITY:
Inclusion Criteria:

* women patients, aged 18-65 years, with an American Society of Anesthesiologists physical status of I or II
* undergoing elective gynaecological laparoscopy for benign diseases

Exclusion Criteria:

* patients who had an allergy or contraindication to any study drug
* had chronic pain or opioid use
* had a history of substance abuse or psychiatric disorders
* were pregnant or lactating
* had a severe cardiovascular, respiratory, renal, hepatic or haematological disease
* had a body mass index >30 kg/m2
* had an inability to understand or cooperate with study procedures

Ages: 33 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale ( VAS ) scores for pain | at 1 hour after surgery
  Pain was assessed at 1 hour to evaluate immediate postoperative pain while allowing time to recover from anaesthesia.
Visual analogue scale ( VAS ) scores for pain | at 2 hours after surgery
  Pain was assessed at 2 hours after surgery.
Visual analogue scale ( VAS ) scores for pain | at 4 hours after surgery
  Pain was assessed at 4 hours after surgery.
Visual analogue scale ( VAS ) scores for pain | at 6 hours after surgery
  Pain was assessed at 6 hours after surgery.
Visual analogue scale ( VAS ) scores for pain | at 12 hours after surgery
  Pain was assessed at 12 hours after surgery.
Visual analogue scale ( VAS ) scores for pain | at 24 hours after surgery
  Pain was assessed at 24 hours after surgery.

SECONDARY OUTCOMES:
the total rescue analgesic consumption (mg) | within 24 hours after surgery
  The total rescue analgesic consumption was calculated by adding the amount of morphine delivered by PCA and any supplemental tramadol given by the nurse for inadequate pain control (VAS >4) or at the patient's request, ensuring that the total opioid dose was within safe limits.
the incidence of postoperative nausea and vomiting(PONV) | within 24 hours after surgery
  The incidence of postoperative nausea and vomiting(PONV) was defined as any nausea, vomiting or both
the nausea severity of postoperative nausea and vomiting(PONV) | within 24 hours after surgery
  The nausea severity was rated on a 4-point scale (0 = none, 1 = mild, 2 = moderate and 3 = severe)
patient satisfaction score | at 24 hours after surgery
  Patient satisfaction was assessed using a 5-point scale (1 = very dissatisfied, 2 = dissatisfied, 3 = neutral, 4 = satisfied and 5 = very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Children's hospital, Wuhan, China